CLINICAL TRIAL: NCT05970393
Title: Inspiratory Contribution of Pressure Support-ventilated Patients in Different PMI Conditions - a Prospective Physiological Study
Brief Title: Inspiratory Contribution of Pressure Support-ventilated Patients in Different PMI Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KY2023-001-02
Record Dates: First submitted 2023-07-01; First posted 2023-08-01 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation
Keywords: pressure support ventilation; inspiratory effort; inspiratory muscle pressure index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): PMI represents the difference between plateau airway pressure and peak airway pressure (plateau - peak) during an end-inspiratory airway occlusion.
  Interventions: Procedure: pressure support level tatrition

INTERVENTIONS:
Procedure: pressure support level tatrition — Baseline ventilators were set by the principle of keeping VT/PBW at 6-8ml/kg and RR at 20-30 breaths/min and the decision of the responsible ICU physician. After then the fraction of inspired oxygen (FiO2), positive expiratory end pressure (PEEP), trigger sensitivity, and cycle-off criteria remain unchanged. Upward and downward PS level adjustments were performed from the baseline PS level at a 1cm H2O interval. Every PS level was maintained for 20 minutes and then three end-inspiratory holdings (2-3seconds) and three end-expiratory holdings were performed. PMI mean value was measured and calculated at every PS level. To avoid additional injury to the lung and diaphragm, the airway peak pressure (Ppeak) was limited to 30cmH2O, and titrating PS was stopped until PMI was less than -1cmH2O and more than 3cmH2O.The inspiratory effort is measured as the pressure generated by inspiratory muscles using esophageal pressure monitoring.

SUMMARY:
Pressure support ventilation (PSV) is an assisted mechanical ventilation mode that provides synchronous inspiratory support for patients with spontaneous breathing. PSV divides the work involved in producing ventilation between the ventilator and the patients. The patient inspiratory effort needs close monitoring to avoid inappropriate assistance and maintain favorable patient-ventilator interaction during PSV. Esophageal pressure (Pes)-derived parameters are regarded as golden indicators of inspiratory effort. Based on this precondition, the fraction of PTP generated by the patient during PSV (PTP ratio) can evaluate the inspiratory contribution proportion of ventilated patients with spontaneous breathing. Inspiratory muscle pressure index (PMI) was confirmed to be associated with inspiratory effort and can effectively predict low/high effort. The study tries to explore the relationship between PMI and PTP ratio and find the optimal cut-off value of PMI to predict different PTP ratios. Second, investigators want to verify the safety and validity of PMI-guided PS settings for pressure-support ventilated patients.

DETAILED DESCRIPTION:
Pressure support ventilation (PSV) is an assisted mechanical ventilation mode that provides synchronous inspiratory support for patients with spontaneous breathing. PSV divides the work involved in producing ventilation between the ventilator and the patients. The level of support should be adjusted to the patient's inspiratory effort for assisted ventilation to be successful. Despite PSV being commonly used in mechanical ventilation therapy, the PS setting is not precisely regulated. Clinicians and respiratory therapists typically use tidal volume/predicted body weight (VT/PBW, 6-8 ml/Kg) and respiratory rate (RR, 20-30 breaths/min) to modify ventilator settings. Because pressure support level is not dynamically modulated based on the inspiratory effort of ventilated patients in time, there is always the risk of excessive or insufficient assistance. Excessive assistance and low inspiratory effort may result in diaphragm disuse atrophy and ventilator-induced lung injury (VILI). Inadequate assistance and high inspiratory effort may result in diagram stretched injury and patient-inflicted lung injury (PSILI). Both situations cause strain and stress on the lung and diaphragm, which may influence the ICU clinical outcomes.

The patient inspiratory effort needs close monitoring to avoid inappropriate assistance and maintain favorable patient-ventilator interaction during PSV. Esophageal pressure (Pes)-derived parameters are regarded as golden indicators of inspiratory effort, including respiratory muscle pressure (Pmus), esophageal pressure-time product (PTPes), etc. Based on this precondition, the fraction of PTP generated by the patient during PSV (PTP ratio) can evaluate the inspiratory contribution proportion of ventilated patients with spontaneous breathing. Pmus index (PMI) is defined as the change in airway pressure (Paw) during the end-inspiratory occlusion and represents the patient's current elastic workload. This variable was confirmed to be associated with inspiratory effort and can effectively predict low/high effort. More importantly, it is non-invasive and available at the bedside because respiratory hold operations are integrated into most ventilators. However, the relationship between PMI and the inspiratory contribution proportion of ventilated patients is not clear, and how to guide PS settings through PMI needs more research.

Our study aims to explore the inspiratory contribution of pressure-support ventilated patients in different PMI conditions. In other words, investigators try to explore the relationship between PMI and PTP ratio and find the optimal cut-off value of PMI to predict different PTP ratios. Second, investigators want to verify the safety and validity of PMI-guided PS settings for pressure-support ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

Adult acute respiratory failure patients undergoing mechanical ventilation were screened daily and enrolled 24 hours after switching to PSV mode.

Exclusion Criteria:

1. age younger than 18 years old and more than 80 years old
2. chronic occlusive pulmonary diseases
3. known pregnancy and parturient
4. gastric, esophageal, and diaphragm surgery
5. barotrauma
6. neuromuscular diseases
7. intracranial hypertension and brain stem injury
8. consciousness level decreased (SAS less than 3 scores)
9. Anticipating withdrawal of life support and/or shift to palliation as the goal of care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The correlation between PMI and PTP ratio | 3 hours
  Regression was conducted by the linear mixed-effects model with patients managed as random effects. The correlation between PMI and PTP ratio was evaluated as the coefficient of determination (R2).
The ability of PMI to detect different PTP ratios | 3 hours
  The ability of PMI to detect different inspiratory effort contribution proportions was assessed using the Area Under the Receiver-Operating-Characteristics Curve (AUROC). The optimal cut-off values were selected based on the Youden index.

SECONDARY OUTCOMES:
Tidal volume per predicted body weight (VT/PBW, ml/Kg) | 3 hours
  We use the VT/PBW (ml/Kg) as lung-protective ventilation safety makers.
Respiratory rate (RR, circle/min) | 3 hours
  We use the RR (circle/min) as lung-protective ventilation safety makers.
Transpulmonary driving pressure (DPlung, cmH2O) | 3 hours
  We use the DPlung (cmH2O) as lung-protective ventilation safety makers.
Respiratory driving pressure (DPrs, cmH2O) | 3 hours
  We use the DPrs (cmH2O) as lung-protective ventilation safety makers.
Respiratory muscle pressure (Pmus, cmH2O) | 3 hours
  Our study chose Pmus (cmH2O) as the golden standard of inspiratory effort to estimate the validity of PMI-guided PS setting.
Esophageal pressure-time product (PTPes, cmH2O) | 3 hours
  Our study chose PTPes (cmH2O) as the golden standard of inspiratory effort to estimate the validity of PMI-guided PS setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao R, Zhou JX, Yang YL, Xu SS, Zhou YM, Zhang L, Miao MY. Use of pressure muscle index to predict the contribution of patient's inspiratory effort during pressure support ventilation: a prospective physiological study. Front Med (Lausanne). 2024 Apr 26;11:1390878. doi: 10.3389/fmed.2024.1390878. eCollection 2024. PMID 38737762